CLINICAL TRIAL: NCT00362934
Title: A Multicenter, Double-Blind, Randomized, Forced-Titration Study to Compare the Efficacy and Safety of the Combination of 145 mg Fenofibrate and 20 or 40 mg Simvastatin With Atorvastatin Monotherapy in Patients With Mixed Dyslipidemia at Risk of Cardiovascular Disease Not Adequately Controlled by 10 mg Atorvastatin Alone
Brief Title: Comparison of the Combination of Fenofibrate and Simvastatin Versus Atorvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Martine Guy, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C LF0242780-01 05 03; 2006-000519-21
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia Combined; efficacy combination fenofibrate simvastatin versus atorvastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — Fenofibrate; Simvastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: fenofibrate / simvastatin
- 2 (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: fenofibrate / simvastatin — Combination of fenofibrate and simvastatin 20 mg and 40 mg
  Arms: 1
Drug: Atorvastatin — Atorvastatin 10 mg and 20mg
  Arms: 2

SUMMARY:
Mixed or combined hyperlipidemia is a common metabolic disorder characterized by both hypercholesterolemia and hypertriglyceridemia. Statins and fibrates have complementary mechanisms and can be coadministered to patients with mixed hyperlipidemia. The overall objective of the study is to compare the efficacy and safety of combining fenofibrate and simvastatin versus atorvastatin monotherapy in patients with mixed hyperlipidemia at risk of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dyslipidemia.

Exclusion Criteria:

* Known hypersensitivity to fenofibrates or simvastatin or atorvastatin
* Pregnant or lactating women
* Contra-indication to fenofibrate or simvastatin or atorvastatin
* Unstable or severe cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 12 weeks of treatment in Triglycerides | 12 weeks
Percent change from baseline to 12 weeks of treatment in HDL-C | 12 weeks
Percent change from baseline to 12 weeks of treatment in LDL-C | 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline to 12 weeks of treatment in Triglycerides | 24 weeks
Percent change from baseline to 12 weeks of treatment in HDL-C | 24 weeks
Percent change from baseline to 12 weeks of treatment in LDL-C | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (68):
- Bulgaria (12):
  - Site 501, Haskovo
  - Site 505, Pleven
  - Site 503, Plovdiv
  - Site 506, Plovdiv
  - Site 500, Sofia
  - Site 502, Sofia
  - Site 504, Sofia
  - Site 507, Sofia
  - Site 509, Sofia
  - Site 511, Sofia
  - Site 508, Varna
  - Site 510, Varna
- Czechia (17):
  - Site 109, Chrudim
  - Site 117, Havířov
  - Site 101, Olomouc
  - Site 114, Olomouc
  - Site 116, Ostrava
  - Site 107, Pardubice
  - Site 111, Pardubice
  - Site 113, Pilsen
  - Site 100, Prague
  - Site 104, Prague
  - Site 108, Prague
  - Site 110, Prague
  - Site 115, Prague
  - Site 103, Teplice
  - Site 106, Trutnov
  - Site 118, Uničov
  - Site 102, Ústí nad Orlicí
- Germany (10):
  - Site 203, Berlin
  - Site 204, Bochum
  - Site 205, Dresden
  - Site 206, Görlitz
  - Site 202, Hamburg
  - Site 208, Karlsruhe
  - Site 207, Leipzig
  - Site 201, Magdeburg
  - Site 209, Nuremberg
  - Site 200, Unterschneidheim
- Slovakia (13):
  - Site 301, Banská Bystrica
  - Site 307, Bratislava
  - Site 310, Bratislava
  - Site 311, Bratislava
  - Site 312, Bratislava
  - Site 309, Dolný Kubín
  - Site 302, Košice
  - Site 305, Lučenec
  - Site 306, Nitra
  - Site 304, Nové Zámky
  - Site 308, Prešov
  - Site 303, Vráble
  - Site 300, Žilina
- Ukraine (16):
  - Site 416, Donetsk
  - Site 401, Kharkiv
  - Site 412, Kiev
  - Site 402, Kyiv
  - Site 404, Kyiv
  - Site 408, Kyiv
  - Site 410, Kyiv
  - Site 414, Lutsk
  - Site 406, Lviv
  - Site 407, Odesa
  - Site 409, Odesa
  - Site 411, Odesa
  - Site 405, Simferopol
  - Site 413, Uzhhorod
  - Site 400, Vinnitsa
  - Site 415, Zaporizhzhya